CLINICAL TRIAL: NCT01618084
Title: A Prospective Randomised Rontgen Stereophotogrammatic Analysis (RSA) Study Using the Uncemented Trident Tritanium Acetabular Component and the Uncemented HA Coated Symax Hip Stem in a Single Centre: Assessment of Implant Migration, Bone Remodeling and Clinical Function
Brief Title: RSA Study Using Two Types of Uncemented Acetabular Components and the Uncemented HA Coated Symax Stem
Acronym: RSA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC10-1-068; NL 33832.068.10 (Other: CCMO)
Record Dates: First submitted 2012-05-22; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis
Keywords: hipreplacement; uncemented; migration; boneremodeling
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tritanium cup (Experimental)
  Interventions: Device: Tritanium acetabular component
- Trident HA cup (Active Comparator)
  Interventions: Device: Tritanium acetabular component

INTERVENTIONS:
Device: Tritanium acetabular component — Total hip arthroplasty using a tritanium uncemented acetabular component

SUMMARY:
The Trident Tritanium acetabular component of a total hip prosthesis is a new developed uncemented acetabular component. In this randomized controlled trial (RCT) the tritanium cup will be compared with the Trident HA acetabular component in two equal sized groups. The Symax HA coated stem will be used as femoral component in both groups.

Study Objectives:

* The primary objective is to determine the prosthetic migration of the uncemented acetabular and femoral total hip components using model based RSA technique
* Secondary objectives are on one hand to assess clinical outcome on the other hand assessing patient satisfaction in both groups using Harris Hip Score, Oxford Hip Score, WOMAC, and EQ-5D questionnaires
* Tertiary objective is to assess bone remodeling of the uncemented acetabular components and the HA-coated Symax hip stem using QCT derived from usinf F18-fluoride PET in a cohort of 12 consecutive patients of this RCT

A total of 50 patients will be enrolled in this RCT divided into two equal groups. Patients have to fulfill the inclusion and exclusion criteria.

All evaluations will be done pre-operatively with 2 weeks before surgery, and after surgery at 4 weeks, 3 and 6 months and 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a BMI < 35
* Patients requiring uncemented primary THA
* Primary diagnosis of osteoarthritis

Exclusion Criteria:

* patients with acetabular or femoral osteotomy
* Patients who had a THA on the contralateral side within last 6 months
* Female patients who are pregnant or planning pregnancy during the course of the study
* Patients with active or suspected infection
* patients with malignancy
* patients with a systemic disease that would effect the subject's welfare or overall outcome of the study
* Patients with a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device
* Patients with systemic or metabolic disorders leading to progressive bone deterioration
* Patients with other illnesses which are likely to affect their outcome
* Patients with known sensitivity to device materials

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
prosthetic migration of the uncemented acetabular and femoral total hip components | 2 years
  determine the prosthetic migration of the uncemented acetabular and femoral total hip components using model based RSA technique

SECONDARY OUTCOMES:
clinical outcome and patient satisfaction | 2 years
  assess clinical outcome and patient satisfaction in both groups using Harris Hip Score, Oxford Hip Score, WOMAC, and EQ-5D questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Lodewijk Van Rhijn, professor, Principal Investigator — Maastricht University Medical centre
Locations (1):
- Maastricht UMC, Maastricht, Netherlands